CLINICAL TRIAL: NCT02856958
Title: Acute Nerve Decompression Versus Non-operative Treatment for Peroneal Nerve Palsy Following Primary Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16041403
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Peroneal Palsy (Foot Drop)
MeSH Terms: conditions — Peroneal Neuropathies

ARMS (2):
- Operative (Experimental): Peroneal nerve decompression
  Interventions: Procedure: Nerve decompression
- Non-operative (Active Comparator): Physical therapy
  Interventions: Other: Non-operative

INTERVENTIONS:
Procedure: Nerve decompression
  Arms: Operative
Other: Non-operative — Physical therapy
  Arms: Non-operative

SUMMARY:
The purpose of this study is to compare acute nerve decompression versus nonoperative treatment in the management of peroneal nerve palsy after total knee arthroplasty (TKA). We hypothesize that acute nerve decompression patients will have better long-term outcomes to patients treated non-operatively for peroneal nerve palsies after TKA.

DETAILED DESCRIPTION:
Peroneal nerve palsy after TKA has been reported in the literature to be 0.3% to 1.5%, although it can be as high as 9.5%. Several risk factors have been described: preoperative valgus deformity and flexion contracture, prolonged intraoperative use of a tourniquet, use of epidural anesthesia, and rheumatoid arthritis. Peroneal palsy is rarely diagnosed on postoperative day 0, but in more than 85% of cases, it presents prior to postoperative day 4.Initial treatment should include flexing the knee, removing any compressive bandages, and discontinuing epidural anesthesia. When there are residual deficits, supportive measures are initiated, including application of an ankle-foot orthosis and physical therapy to prevent ankle contracture. If there is no clinical recovery by six to twelve weeks, electromyography (EMG) is typically performed. Some clinicians have advocated the use of EMG studies in the acute phase. In cases of incomplete recovery, delayed surgical exploration and decompression of the peroneal nerve is an option that has been reported to improve outcomes. Unfortunately, not all cases respond, even with surgical treatment. In addition, little information is available describing the outcomes of acute surgical decompression for peroneal nerve palsy after total knee arthroplasty.

While there have been retrospective case reports and series that have examined outcomes after delayed peroneal nerve decompression, we are unaware of reports describing acute decompression. Delayed decompression of the peroneal nerve has been associated with the return of nerve function. Krackow et al. reported the results of five patients who underwent delayed surgical decompression for peroneal nerve palsy after total knee arthroplasty at an average of 27.2 months (range, 5-50 months) and found that 100% were able to discontinue use of the ankle-foot orthosis and 80% had full neurological recovery. The patient who had partial return of neurological function did not undergo decompression until almost four years postoperatively. Mont et al. found that, in patients who underwent surgical peroneal nerve decompression two to sixty months following total knee arthroplasty, 97% reported functional and subjective improvements at a mean of three years post-decompression and were able to discontinue use of the ankle-foot orthosis. Only 33% of the patients who were managed nonoperatively reported improvement in functional and subjective outcomes.

Therefore, in 33% of the patients, an acute decompression would not have been necessary, but in the other 67%, it may have been beneficial. In both studies, patients underwent a trial of nonoperative treatment, and no patient underwent a peroneal nerve decompression earlier than two months after the index total knee arthroplasty. Initial experience with two peroneal nerve palsies following TKA has encouraged some institutions to offer acute decompression to all patients who present with peroneal palsy following total knee arthroplasty. This parallels the practice patterns regarding the wrist, where an acute carpal tunnel release is performed to avoid complications when a patient demonstrates carpal tunnel compressive symptoms postoperatively from wrist surgery. While most patients will improve with nonoperative treatment over time, acute decompression may accelerate recovery, which can decrease uncertainty and stress for both the patient and the surgeon. The surgical technique is relatively straightforward; however, the surgeon and patient must consider the risks of a second anesthetic and operation. In previous experiences with both acute and delayed decompression, while direct damage to the nerve itself is rare, fascial bands, hematomas, and local edema are typically identified that contribute to the compression of the peroneal nerve. Therefore, while nonoperative treatment would possibly result in a return of nerve function once the hematoma resorbed and edema decreased, there may still be some residual dysfunction from the time period of nerve compression and thickened fascial bands around the nerve. Additional study of acute decompression is warranted to understand if it offers both short and long-term advantages over nonoperative treatment.

Treatment Groups: Acute Nerve Decompression - patients will initially receive conservative management (flexing the knee, removing any compressive bandages, and discontinuing epidural anesthesia) followed by a peroneal nerve decompression within 1 week of diagnosis of peroneal nerve palsy. Decompression involves surgical intervention in the setting of a sterile operating room. The patient will be provided with multiple options of anesthesia (per discussion with the anesthesia team). The surgical procedure involves an incision at the lateral aspect of the knee, near the proximal fibula at the level of the fibular neck. The peroneal nerve is carefully identified and dissected. Tissue surrounding or impinging the nerve is carefully removed or cut to rid the compressive environment. The nerve is re- examined to ensure there are no additional points of compression/irritation. The soft-tissues and skin are subsequently closed with suture. Nonoperative Treatment - patients will receive conservative management (flexing the knee, removing any compressive bandages, and discontinuing epidural anesthesia) as well as supportive measures (ankle-foot orthosis and physical therapy) for symptoms lasting longer than 6 week. Outcome Measures: Primary Measure - ≥ 3/5 dorsiflexion strength 3 months after surgery/randomization

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting with peroneal palsy (< 3/5 dorsiflexion) within 3-weeks after primary TKA

Exclusion Criteria:

* Patient's with pre-existing peroneal palsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Dorsiflexion strength | within 3 months from surgery

CONTACTS AND LOCATIONS:
Overall Officials: John J Fernandez, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Midwest Orthopedics at Rush, Chicago, Illinois, United States